CLINICAL TRIAL: NCT01884090
Title: Youth Empowerment Solutions for Positive Youth Development (YES) Also Known as Genesee County Afterschool Study (GCAS)
Brief Title: Youth Empowerment Solutions for Positive Youth Development
Acronym: YES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Marc A. Zimmerman, Professor, Department of Health Behavior and Health Education, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R01HD062565 (NIH)
Record Dates: First submitted 2012-10-23; First posted 2013-06-21 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Violence; Child or Adolescent Antisocial Behavior
Keywords: Empowerment; Youth; Violence; Community; Prevention
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Youth Empowerment Solutions (YES) (Experimental): Participants receiving the The 16-week, 30-session YES curriculum YES as a part of the 21st Century after-school program at middle schools that have high economic and academic needs. 21st Century is a U.S. Department of Education program which provides academic enrichment opportunities during non-school hours and during the summer for children who attend low-performing schools in areas with high poverty (U.S. Department of Education, 2009).
  Interventions: Behavioral: Youth Empowerment Solutions (YES)
- Standard After School Programming (Active Comparator): Youth in the comparison arm of the study will participate in standard after-school programming administered by Flint Community Schools and Genesee Intermediate School District. The standard program is the 21st Century after-school program at middle schools that have high economic and academic needs. 21st Century is a U.S. Department of Education program which provides academic enrichment opportunities during non-school hours and during the summer for children who attend low-performing schools in areas with high poverty (U.S. Department of Education, 2009)
  Interventions: Behavioral: Youth Empowerment Solutions (YES)

INTERVENTIONS:
Behavioral: Youth Empowerment Solutions (YES) — Participants receiving the The 16-week, 30-session YES curriculum YES as a part of the 21st Century after-school program at middle schools that have high economic and academic needs. 21st Century is a U.S. Department of Education program which provides academic enrichment opportunities during non-school hours and during the summer for children who attend low-performing schools in areas with high poverty (U.S. Department of Education, 2009).
  Other Names: Genesee County Afterschool Study

SUMMARY:
The Youth Empowerment Solutions for Positive Youth Development (YES) Study , is a randomized controlled trial that compares youth in standard after school programs offering activity choice (e.g. sports, academic enrichment, arts) to youth assigned to an after school program that includes training in community development, formation of intergenerational partnerships and experience conducting community improvement projects. The study aims are to: 1) implement and evaluate an empirically developed intervention for empowering youth (YES) using a randomized controlled trial design in a high risk urban and suburban sample; 2) test a conceptual model that posits a causal relationship from youth empowerment processes to positive developmental outcomes; and 3) follow youth over time to assess sustainability of gains in healthy development. Developmental outcomes will be assessed at baseline, curriculum completion and at three and nine months post-intervention.

This study will be referred to as the Genesee County Afterschool Study (GCAS) in recruitment, consents, assents and promotional materials. The study compares different types of after school programs, and we will be randomly assigning students into two groups, 1) the "regular" 21st Century Afterschool programs and 2) the "regular" 21st Century Afterschool programs with the YES supplement. We do not want to bias desirability of the random groups by naming one of the groups to be tested in the study name. Therefore, in documents we will refer to the study as the "Genesee County Afterschool Study (GCAS)."

Study hypotheses:

1. Youth in the YES intervention arm will demonstrate increased intrapersonal, interactional, and behavioral empowerment than youth in the comparison group arm.
2. Youth in the YES intervention arm will demonstrate higher scores on the positive developmental outcome variables, and lower scores on the negative developmental outcome variables, than youth in the comparison group arm.
3. Behavioral empowerment will partially mediate the relations between intrapersonal and interactional empowerment and youth developmental outcomes, such that youth with greater intrapersonal and interactional empowerment skills will demonstrate increased behavioral empowerment, which in turn will result in higher scores on positive developmental outcome variables, and lower scores on negative developmental outcome variables.

DETAILED DESCRIPTION:
YES is a partnership between the University of Michigan School of Public Health, the Flint Community Schools and the Genesee County Intermediate School District. The study will include participants at eight high-need middle schools with 21st Century after school programs.

Researchers have consistently found that participation in out of school programs enhances adolescents' well being and sense of worth, involves them in positive behaviors and helps them avoid involvement in problem behaviors. Although key elements of successful after school programs have been proposed (e.g., adult mentorship), the processes through which youth positive outcomes are achieved have rarely been empirically examined. Empowerment theory provides a unique conceptual framework for developing programs to enhance positive youth development because it incorporates the notion that health promotion requires not only that youth develop specific skills and positive assets, but also that youth become motivated to actively apply these skills and knowledge to become agents of positive change for themselves and in their communities. Thus, programs based on empowerment theory focus on building positive assets, connecting youth with local resources and adult role models, and engaging youth in community service activities. Ecological theory complements empowerment theory because it focuses attention on the social contexts in which youth develop, interactions between these contexts, and the roles youth can play in these contexts (e.g., schools, communities). An intervention approach informed by these two theories should enhance positive youth development by engaging youth in relevant ecological settings where they can learn skills, practice those skills, and establish the social resources to effectively navigate the social contexts in which they find themselves and develop into healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Students entering 7th grade
* Students enrolled enrolled in the 21st Century After School Program at eight middle schools in Genesee County, Michigan

Exclusion Criteria:

* None

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 418 (Actual)
Dates: Start 2011-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Intrapersonal Empowerment | 1 year
  Scales will include Self-Acceptance, Mastery, Leadership Efficacy, and Motivation to Control.
Interactional Empowerment | 1 year
  Scales will include Adult Mentoring Relationships, Adult Resources, and Resource Mobilization.
Behavioral Empowerment | 1 year
  Scales will include Leadership Behavior, Community Engagement, and School Engagement

SECONDARY OUTCOMES:
School Bonding | 1 year
  Scales include: school engagement; social support from teachers and staff
Academic Achievement | 1 year
  Scales include: academic effort and achievement. Will track participants grades.
Social Competence | 1 year
  Scales include: social skills rating; responsible decision-making
Prosocial Activities | 1 year
  Scales include: participation in extracurricular activities, pro-social scale
Antisocial Behavior | 1 year
  scales include: anti-social attitudes and behavior, attitude toward conflict; beliefs supporting aggression, perpetration of aggression, rule-breaking behavior
Substance Use | 1 year
  Scale includes 8 items from National Survey on Drug Use and Health
Internalizing Problems | 1 year
  Scales include: anxiety, depression

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Zimmerman, PhD, Principal Investigator — University of Michigan
Locations (11):
- United States (11):
  - Bentley Schools, Burton, Michigan
  - Atherton Middle School, Burton, Michigan
  - Bendle Middle School, Burton, Michigan
  - Hamady Middle School, Flint, Michigan
  - Northern High School, Flint, Michigan
  - Northwestern High School, Flint, Michigan
  - Kearsley Schools, Flint, Michigan
  - Carman-Ainsworth Middle School, Flint, Michigan
  - Genesee School District, Genesee, Michigan
  - Beecher Middle School, Mt. Morris, Michigan
  - Mt. Morris Junior High, Mt. Morris, Michigan

REFERENCES:
- [Background] Zimmerman MA, Stewart SE, Morrel-Samuels S, Franzen S, Reischl TM. Youth Empowerment Solutions for Peaceful Communities: combining theory and practice in a community-level violence prevention curriculum. Health Promot Pract. 2011 May;12(3):425-39. doi: 10.1177/1524839909357316. Epub 2010 Nov 8. PMID 21059871
- [Background] Franzen S, Morrel-Samuels S, Reischl TM, Zimmerman MA. Using process evaluation to strengthen intergenerational partnerships in the Youth Empowerment Solutions program. J Prev Interv Community. 2009;37(4):289-301. doi: 10.1080/10852350903196290. PMID 19830624
- [Background] Griffith DM, Allen JO, Zimmerman MA, Morrel-Samuels S, Reischl TM, Cohen SE, Campbell KA. Organizational empowerment in community mobilization to address youth violence. Am J Prev Med. 2008 Mar;34(3 Suppl):S89-99. doi: 10.1016/j.amepre.2007.12.015. PMID 18267207
- [Background] Reischl TM, Zimmerman MA, Morrel-Samuels S, Franzen SP, Faulk M, Eisman AB, Roberts E. Youth empowerment solutions for violence prevention. Adolesc Med State Art Rev. 2011 Dec;22(3):581-600, xiii. PMID 22423465
- [Background] Eisman AB, Zimmerman MA, Kruger D, Reischl TM, Miller AL, Franzen SP, Morrel-Samuels S. Psychological Empowerment Among Urban Youth: Measurement Model and Associations with Youth Outcomes. Am J Community Psychol. 2016 Dec;58(3-4):410-421. doi: 10.1002/ajcp.12094. Epub 2016 Oct 6. PMID 27709632
- See also: Youth Empowerment Solutions homepage — http://yes.sph.umich.edu/